CLINICAL TRIAL: NCT02145078
Title: A Pilot Trial of Platinum, Gemcitabine, or Pemetrexed Single- or Multi-Agent Therapy With Serial Tumor Specimen Collection in Patients With Advanced Non-Small-Cell Lung Cancer
Brief Title: Gene Expression Levels in Predicting Treatment Response in Patients With Stage IV Non-small Cell Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Gerold Bepler, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-177; NCI-2014-01023 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1402012854; 2013-177 (Other: Barbara Ann Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Pemetrexed; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy regimen) (Experimental): Patients receive 1 of 4 chemotherapy regimens at the discretion of the primary oncologist following institutional guidelines, including cisplatin, carboplatin, pemetrexed disodium IV on day 1, or gemcitabine hydrochloride IV on days 1 and 8. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. After course 2, patients may continue treatment off-study at the discretion of the treating physician.
  Interventions: Drug: docetaxel; Drug: pemetrexed disodium; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Drug: pemetrexed disodium — Given IV
  Other Names: ALIMTA; LY231514; MTA
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies whether the levels of certain genes in the tissue and blood are related to how well patients with stage IV non-small cell lung cancer respond to chemotherapy. Genes may affect how sensitive or resistant tumors are to chemotherapy. Studying the levels of genes related to tumor response before and after chemotherapy may help doctors learn whether they can predict how well patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the association between baseline gene expression levels at the protein and messenger ribonucleic acid (mRNA) level and best treatment response after two cycles of single-agent or multi-agent chemotherapy

SECONDARY OBJECTIVES:

I. To describe changes in protein and mRNA levels of ribonucleotide reductase M1 (RRM1), thymidylate synthetase (TS), and excision repair cross-complementing rodent repair deficiency, complementation group 1 (ERCC1) in serial biopsies obtained from patients being treated with gemcitabine (gemcitabine hydrochloride), pemetrexed (pemetrexed disodium), and platinum.

II. To describe the association between changes in marker levels and changes in tumor diameters.

TERTIARY OBJECTIVES:

I. To explore the relationship between marker levels in circulating tumor cells and solid tumor specimens.

II. To explore the relationship between marker levels in viable peripheral blood mononuclear cells (PBMCs), circulating tumor cells, and tumor specimens.

III. Should sufficient amounts and numbers of tumor specimens remain after these analyses, they will be used to assess if other genes implicated in non-small cell lung cancer (NSCLC) outcome and response to treatment might be useful as prognostic or predictive markers for patient outcome.

OUTLINE:

Patients receive 1 of 3 chemotherapy regimens at the discretion of the primary oncologist, including docetaxel intravenously (IV) on day 1, pemetrexed disodium IV on day 1, or gemcitabine hydrochloride IV on days 1 and 8. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. After course 2, patients may continue treatment off-study at the discretion of the treating physician.

After completion of study treatment, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced stage NSCLC who are candidates for single or multi-agent first-line therapy.
* Second-line or higher therapy for any patients with NSCLC with performance status (PS) 0-2
* Maintenance therapy for patients after completion of four cycles of dual-agent platinum-based chemotherapy
* Stage IV, histologically or cytologically confirmed NSCLC; confirmation may be obtained with the first protocol-specified tumor biopsy
* White blood cell count > 3000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 9.0 g/dl
* A tumor lesion that can be safely biopsied as judged by the treating oncologist and physician performing the procedure and has not been radiated
* At least one unidimensionally measurable tumor lesion >= 1 cm in longest diameter using spiral CT (>= 2 cm in longest diameter by any other technique) that has not been radiated and is not located in a bone
* Performance status 0-2 by Eastern Cooperative Oncology Group criteria
* Life expectancy of >= 3 months
* Able to understand and sign the informed consent document

Exclusion Criteria:

* Therapy that does not include cisplatin, carboplatin, gemcitabine, and/or pemetrexed
* Concomitant medical or psychiatric illness that is likely to interfere with a reasonably safe execution of the treatment plan
* Concomitant malignancy other than NSCLC that requires active therapy; prior malignancies are allowed as long as the disease is controlled and does not require ongoing therapy of any kind; prior therapy must have concluded at least 1 year before treatment initiation on this protocol; exceptions are non-melanoma skin cancer, prostate cancer and prostatic intraepithelial neoplasia (PIN) treated with local intervention and deemed cured, cervical cancer and carcinoma in situ (CIS) treated with local intervention and deemed cured, and laryngeal cancer and CIS treated with local intervention and deemed cured
* Carcinomatous meningitis
* Uncontrolled central nervous system (CNS) disease
* The time interval between CNS radiation, whole brain radiation, spinal cord radiation, or radiosurgery, and initiation of protocol specified chemotherapy must be at least 1 week
* Malignant pleural, pericardial, or peritoneal effusion if it is the only site of disease activity; i.e., if no other measurable tumor lesions exist
* Coagulopathy or anticoagulation therapy that cannot be safely corrected or interrupted for tumor biopsy
* Significant hepatic dysfunction, renal dysfunction, or metabolic derangement that precludes full-dose chemotherapy at the specified starting doses
* Concomitant treatment with chemotherapeutic agents for diseases other than malignancy
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06-18 (Actual); Study Completion 2017-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerold Bepler, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemotherapy Regimen)
Started | 4
Completed | 0
Not Completed | 4
Not completed — Death | 1
Not completed — Reason not given | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy Regimen)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 62 [50 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Baseline Marker Measurement
Description: A univariable regression of continuous disease response on baseline marker value will be performed. A multivariable regression model adjusted for clinical covariates will be evaluated as well. Expression levels of RRM1, TS, BRCA1, and other molecules and disease response after course 2 will be log-transformed.
Time Frame: Baseline
Population: No patient was analyzed.
Arm/Group | Treatment (Chemotherapy Regimen)
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Biomarker Expression Levels
Description: Evaluated using Pearson correlation. If data are not normally distributed after log transformation, a non-parametric method (e.g., Spearman correlation) will be used.
Time Frame: Baseline to up to 8 weeks (after course 2)
Population: No patient was analyzed.
Arm/Group | Treatment (Chemotherapy Regimen)
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Since, the study was canceled due to slow accrual, no biomarkers were measured; therefore, no analysis with biomarkers. Only the OS will be calculated.
Time Frame: From the date of protocol-specified treatment initiation to the date of death or last observation, assessed up to 12 months
Population: All eligible patients.Since, the study was canceled due to slow accrual, no biomarkers were measured; therefore, no analysis with biomarkers. Only the OS will be calculated.
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Chemotherapy Regimen)
Number analyzed (Participants) | 4
months | 2.0 [1.1 to 7.0]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Each biomarker evaluated using its expression level (continuous variable) and dichotomous form (based on a median cutoff). A univariable Cox regression model will be used to assess the relationship of expression levels of each biomarker to PFS. In addition, for the dichotomous variables, the sample will be divided into those above and below the median for each biomarker. PFS probabilities for each group will be estimated using the Kaplan-Meier method, with standard errors based on Greenwood's formula. Log rank tests will be used to determine the level of significance between survival curves. Since, the study was canceled due to slow accrual, no biomarkers were measured; therefore, no analysis with biomarkers. Only the PFS will be calculated.
Time Frame: From the date of protocol-specified treatment initiation to the date of progression, death, or last observation, assessed up to 12 months
Population: No analysis with biomarkers.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Chemotherapy Regimen)
Number analyzed (Participants) | 4
days | 42 [34 to 60]

5. Secondary Outcome: Expression Levels of Biomarkers and Other Molecules
Description: To assess the relationship between expression levels of RRM1, TS, BRCA1, and other molecules and demographic and disease variables, the Wilcoxon rank sum test or Kruskal-Wallis test for dichotomous or polychotomous categorical variables (such as sex, and histology) and the Spearman correlation coefficient for continuous ordinal variables (such as age or stage) will be used.
Time Frame: Up to 8 weeks (end of course 2)
Population: No patient was analyzed.
Arm/Group | Treatment (Chemotherapy Regimen)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 months
Description: Only biopsy related AEs and SAEs were to be reported.
Arm/Group | Treatment (Chemotherapy Regimen)
All-Cause Mortality (participants affected / at risk) | 4/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
This study was stopped because of low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT02145078/Prot_SAP_000.pdf